CLINICAL TRIAL: NCT07226323
Title: Testing the WeCare Intervention to Address Mental Health and Medication Adherence Challenges Among MSM in South Africa
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Don Operario, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00009339; 5R34MH135806-02 (NIH); 2025P010078 (Other: Emory IRB)
Record Dates: First submitted 2025-11-07; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: HIV Infections; Mental Health
Keywords: Men having sex with Men; Medication adherence; PrEP Adherence; ART Adherence
MeSH Terms: conditions — HIV Infections; Psychological Well-Being; Medication Adherence | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Friendship Bench (FB) arm (Experimental)
  Interventions: Behavioral: WeCare
- Control Arm (Other)
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: WeCare — The intervention is an adapted Friendship Bench (FB) for MSM in South Africa that integrates counseling on HIV medication adherence and the mental health-adherence relationship. The intervention includes up to 4 individual sessions and up to 4 group sessions; individual sessions may be delivered in person or online (Inuka-style), while all group sessions are in person.
  Arms: Friendship Bench (FB) arm
Behavioral: Standard of Care — The control group will receive enhanced standard care at POP INN Wellness Clinic: psychoeducation for all PrEP/ART enrollees, free medication, access to ongoing support groups, and referrals provided by the clinic.
  Arms: Control Arm

SUMMARY:
The goal of this clinical trial is to learn if the WeCare intervention-an adapted Friendship Bench program that integrates problem-solving therapy, minority-stress-informed content, and explicit PrEP/ART adherence skills-improves mental health and HIV medication adherence among men who have sex with men (MSM). It will also assess the safety, acceptability, and feasibility of delivering WeCare through trained lay coaches in community clinics.

Main questions the trial aims to answer:

* Does WeCare reduce symptoms of depression and anxiety among MSM?
* Does WeCare improve PrEP and ART adherence and increase rates of viral suppression among participants on ART?
* Is WeCare acceptable, feasible, and safe when delivered by lay coaches in POP INN clinics compared with usual care?

DETAILED DESCRIPTION:
Men who have sex with men (MSM) in sub-Saharan Africa face very high HIV incidence and prevalence, with South Africa carrying the largest national burden and an estimated ~30% HIV prevalence among MSM. National policies in South Africa endorse universal test-and-treat and prioritize MSM for Pre-Exposure Prophylaxis (PrEP) and Anti-Retroviral Therapy (ART), but care cascade indicators and adherence outcomes for MSM lag behind national averages, indicating a need for differentiated, targeted service approaches.

Common mental health problems are prevalent among MSM and are strongly associated with poorer PrEP and ART adherence. Randomized and quasi-experimental trials in the region show that lay-delivered or nurse-delivered mental health interventions can reduce depression and improve ART adherence and viral suppression, while observational studies link poor mental health to lower PrEP adherence and limited trial evidence suggests integrated adherence interventions may improve biomarker outcomes.

The Friendship Bench (FB) model-an evidence-based, lay health worker-delivered problem-solving therapy program developed in Zimbabwe and adapted across low-resource settings-produces substantial reductions in depressive symptoms and can be delivered in person or digitally. FB's original form had limited effects on ART adherence, prompting calls to explicitly integrate adherence counseling; systematic adaptation is required to make FB effective for MSM by incorporating minority stress theory, addressing anti-MSM stigma and disclosure challenges, and adding explicit adherence skills training.

Aurum's POP INN clinics provide MSM-friendly services and peer support and have piloted FB-style coaching, revealing high rates of medication adherence challenges and moderate-to-severe depression among MSM. Pilot quantitative and qualitative data identify predictors of non-suppression and adherence problems-such as clinic location, transactional sex, missed doses, anxiety, and shorter ART duration-and show a clear preference among MSM for HIV status-neutral programming. Building on these findings, the proposed WeCare intervention aims to adapt Facebook into a status-neutral, minority-stress-informed package that integrates problem-solving therapy with explicit PrEP/ART adherence support, delivered by trained lay coaches, to improve mental health, medication adherence, viral suppression, stigma reduction, and community cohesion.

ELIGIBILITY:
Inclusion Criteria:

* Male
* reports sexual intercourse with a man in the past 6 months
* reside in the Johannesburg metropolitan area with no plans to relocate during the next 6 months
* ability to communicate in English
* current prescription for any ART regimen (HIV-positive participants) or daily oral PrEP (HIV-negative participants) at the POP INN clinic.
* HIV positive participant only: unsuppressed HIV viral load (HIV-1 RNA viral load ≥200 copies/mL) in the sample collected in the past six months
* HIV negative participants only: Self-reported challenges adhering to daily oral PrEP (i.e miss 3 or more tablets per week)
* Moderate symptoms of depression during past 2 weeks (score on the PHQ-9 ≥10 and <20)
* Ability to understand and provide informed consent.

Exclusion Criteria:

* Presently engaged in mental health therapy.
* Participated in qualitative phase of WeCare study (AUR2-18-419) or open-pilot (present study).
* Refuses audio recording of the in-person or online individual counselling session

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Assessment : Modified version of the Session Evaluation Form (SEF) score | Baseline, Month 3, Month 6
  13-item SEF measuring perceived feasibility, acceptability, and intervention utility.
  Composite scores are calculated with higher scores indicating more perceived feasibility and acceptability.
Change in Client Satisfaction Survey (CSQ-8) score | Baseline, Month 3, Month 6
  8-item CSQ assessing satisfaction with recruitment, retention, and intervention procedures, engagement data from the trial (e.g., completion of sessions).
  Composite scores are calculated with higher scores indicating more satisfaction.
Mental health measures: Change in The Patient Health Questionnaire (PHQ-9) scores | Baseline, Month 3, Month 6
  The Patient Health Questionnaire (PHQ-9) measures the frequency of depression symptoms within the past two weeks. The PHQ-9 comprises five categories, where a cut-off point of 0-4 indicates no depressive symptoms, 5-9 mild depressive symptoms, 10-14 moderate depressive symptoms, 15-19 moderately-severe depressive symptoms, and 20-27 severe depressive symptoms
Change in Psychological stress: WHO Self-Reporting Questionnaire-20 (SRQ-20) score | Baseline, Month 3, Month 6
  The WHO Self-Reporting Questionnaire-20 (SRQ-20) includes items to reflect symptoms of depression, anxiety and psychosomatic complaints, which are all together grouped under the heading of common mental disorder (CMD) and have been found to detect probable mental health disorder with satisfactory accuracy
Change in ART adherence | Baseline, Month 3, Month 6
  ART adherence will be defined as a suppressed HIV viral load (HIV-1 RNA viral load <200 copies/mL) in a blood sample
Change in PrEP adherence | Baseline, Month 3, Month 6
  PrEP adherence will be defined as an intracellular Tenofovir Diphosphate (TFV-DP) concentration ≥700 fmol/punch in a dried blood spot (DBS) sample. This concentration was found consistent with an average of ≥4 doses/week in the prior month in a directly observed study among men and women in the United States

SECONDARY OUTCOMES:
Self reported medication adherence | Baseline, Month 3, Month 6
  Adherence outcomes will be based on self-report data, where participants will be asked, "How many days did you not take your PrEP in the past 30 days (0-30 days)
Status neutral composite adherence | Baseline, Month 3, Month 6
  Based on Tenofovir Diphosphate (TFV-DP) concentration ≥700 fmol/punch OR HIV-1 RNA viral load <200 copies/ml

CONTACTS AND LOCATIONS:
Overall Officials: Don Operario, PhD, Principal Investigator — Rollins School of Public Health
Locations (1):
- Aurum Institute, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with researchers who submit a methodologically sound proposal. Data will be collected by Aurum; Aurum will share de-identified data with Emory (including data dictionaries).
Supporting Information: Study Protocol, ICF
Time Frame: Data will be shared following publication